# STATISTICAL ANALYSIS PLAN Protocol FX006-2019-017

A Single-arm, Open-label Study to Evaluate a Procedure for Intra-articular (IA) Injection of FX006 in Patients with Osteoarthritis (OA) of the Hip

Protocol Number: FX006-2019-017

(Version Date) Version 1.0 (28 June 2019)

Name of Test Drug: FX006

Phase: 2

**Methodology:** Single-arm, open-label study

**Sponsor:** Flexion Therapeutics 10 Mall Road, Suite 301

Burlington, Massachusetts, USA

Tel: 781-305-7777

**Sponsor Representative:** 

Amy Cinar, PhD

Director, Biostatistics

**Document Date:** December 18, 2019

**Document Version:** Version 1.0

### Confidentiality

This document is confidential and proprietary property of Flexion Therapeutics, Inc. and to be used only as authorized by Flexion Therapeutics, Inc.. No part is to be reproduced, disclosed to others, or quoted without prior written authorization from Flexion Therapeutics, Inc.

| SIGNATURE PAGE | |
|---|---|
| Protocol Title: | A Single-arm, Open-label Study to Evaluate a<br>Procedure for Intra-articular (IA) Injection of FX006 in<br>Patients with Osteoarthritis (OA) of the Hip |
| Sponsor: | Flexion Therapeutics<br>10 Mall Road, Suite 301<br>Burlington, Massachusetts, USA<br>Tel:781-305-7777 |
| Protocol Number: | FX006-2019-017<br>Version 1.0 (28 June 2019) |
| <b>Document Title:</b> | Statistical Analysis Plan, Protocol FX006-2019-017 |
| <b>Document Date / Version</b> | 18 December 2019 / Final Version 1.0 |
| Cytel, Inc. Author: | |
| Laurel Bastone | Signature: |
| Associate Director, Biostatistics | |

Date:\_\_\_\_

### **Sponsor Approval**

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol, clinical development plan, and all applicable regulatory guidances and guidelines.

I have discussed any questions I have regarding the contents of this document with the biostatistical author.

**Sponsor Signatories:** 

I also understand that any subsequent changes to the planned statistical analyses, as described herein, may have a regulatory impact and/or result in timeline adjustments. All changes to the planned analyses will be described in the clinical study report (CSR).

# Amy Cinar, PhD Signature: Director, Biostatistics Date: Scott Kelley, MD Signature: Chief Medical Officer

# TABLE OF CONTENTS

| | | Section | Page |
|----|--------|-----------------------------------------------|------|
| 1. | INTR | ODUCTION AND OBJECTIVES OF ANALYSIS | 9 |
| | 1.1. | Introduction | 9 |
| | 1.2. | Objectives of Statistical Analysis | 11 |
| 2. | STUD | OY DESIGN | 12 |
| | 2.1. | Synopsis of Study Design | 12 |
| | 2.2. | Study Procedures | 12 |
| | 2.3. | Efficacy Endpoints | 13 |
| | | 2.3.1. Primary Efficacy Endpoint | 13 |
| 3. | PATI | ENT POPULATIONS | 14 |
| | 3.1. | Population Definitions | 14 |
| 4. | STAT | TISTICAL METHODS | 15 |
| | 4.1. | Sample Size Justification | 15 |
| | 4.2. | General Statistical Methods and Data Handling | 15 |
| | 4.2.1. | General Methods | 15 |
| | 4.2.2. | Computing Environment | 15 |
| | 4.2.3. | Methods of Pooling Data | 16 |
| | 4.2.4. | Adjustments for Covariates | 16 |
| | 4.2.5. | Multiple Comparisons/Multiplicity | 16 |
| | 4.2.6. | Subpopulations | 16 |
| | 4.2.7. | Discontinuations and Loss to Follow-up | 16 |
| | 4.2.8. | Missing, Unused, and Spurious Data | 16 |
| | 4.2.9. | Visit Windows | 16 |
| | 4.2.10 | . Baseline definitions | 17 |
| | 4.3. | Interim Analyses | 17 |
| | 4.4. | Final Analyses | 17 |
| | 4.5. | Patient Disposition | 17 |
| | 4.6. | Protocol Deviations | 17 |
| | 4.7. | Demographic and Baseline Characteristics | 18 |
| | 4.7.1. | Demographic Characteristics | 18 |
| | 4.7.2. | OA Medical History | 18 |

| | | Section | Page |
|----|--------|------------------------------------------------|------|
| | 4.7.3. | Prior medication | 18 |
| | 4.8. | Study Drug Exposure | 19 |
| | 4.9. | Efficacy Evaluation | 19 |
| | 4.10. | Safety Analyses | 19 |
| | | 4.10.1. Adverse Events | 19 |
| | | 4.10.2. Laboratory Data | 21 |
| | | 4.10.3. Vital Signs and Physical Examinations | 21 |
| | | 4.10.4. Index Hip Assessment and Aspiration | 21 |
| | | 4.10.5. Index Hip X-Ray | 21 |
| | | 4.10.6. Concomitant Medications | 22 |
| | | 4.10.7. Surgical Procedures | 22 |
| 5. | CHA | NGES TO PLANNED ANALYSES | 23 |
| 6. | Refer | ences | 24 |
| 7. | CLIN | ICAL STUDY REPORT APPENDICES | 26 |
| | 7.1. | Statistical Tables and Figures to be Generated | 26 |
| | 7.2. | Data Listings to be Generated | 27 |
| | 7.3. | Laboratory Unit Conversion Factors | 29 |
| | 7.4. | Laboratory Normal Ranges | |
| | 7.5. | Laboratory Grade Definitions - CTCAE 4.03 | 38 |

| LIST OF IN | I-TEXT TABLES | |
|------------|-------------------------------|------|
| Table | | Page |
| Table 1 | Schedule of Study Assessments | 13 |

### **ABBREVIATIONS**

| Abbreviation | Definition |
|--------------|----------------------------------------------------|
| AE | Adverse Event |
| ACR | American College of Rheumatology |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| cm | Centimeter |
| CM | Concomitant Medications |
| CMC | Carboxymethylcellulose Sodium |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| eCRF | Electronic Case Report Form |
| EOS | End of Study |
| EULAR | European League Against Rheumatism |
| HDL | High Density Lipoprotein |
| HIV | Human Immunodeficiency Virus |
| IA | Intra-articular |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| JSN | Joint Space Narrowing |
| KL | Kellgren-Lawrence |
| kg | Kilogram |
| LDL | Low Density Lipoprotein |
| LLN | Lower Limit of Normal |
| m | Meter |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| NaCl | Sodium Chloride |
| OA | Osteoarthritis |
| OARSI | Osteoarthritis Research Society International |
| PDF | Portable Document Format |
| Ph. Eur/USP | Pharmacopoeia Europaea/ United States Pharmacopeia |
| PLGA | Poly (Lactic-co-Glycolic Acid) |
| PT | Preferred Term |
| SAE | Serious Adverse Event |

| Abbreviation | Definition |
|--------------|---------------------------|
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SP | Safety Population |
| TA | Triamcinolone Acetonide |
| TEAE | Treatment Emergent AE |
| ULN | Upper Limit of Normal |
| US | United States |
| WHO | World Health Organization |

<sup>&</sup>lt;sup>1</sup> Abbreviated in past protocols and documents as TCA

### 1. INTRODUCTION AND OBJECTIVES OF ANALYSIS

### 1.1. Introduction

Osteoarthritis (OA) is a painful and debilitating musculoskeletal disease that is characterized by intraarticular (IA) inflammation, deterioration of articular cartilage, and degenerative changes to peri-articular and subchondral bone (Creamer and Hochberg, 1997; Goldring and Goldring, 2006). Arthritis is the most common cause of disability in the United States of America (USA), and OA is the most common joint disease, affecting 31 million Americans, with numbers expected to grow as a result of aging, obesity and sports injuries (Cisternas et al., 2016). Recent data suggest that OA accounts for over \$185 billion of annual healthcare expenditures in the US, which does not include loss of productivity costs. It is estimated that by 2030, 45 million people will have OA. OA commonly affect large weight-bearing joints like the knees and hips, but also occurs in the shoulders, hands, feet and spine. Patients with OA suffer from joint pain, tenderness, stiffness and limited movement. As the disease progresses, it becomes increasingly painful and debilitating, culminating, in many cases, in the need for total joint arthroplasty.

Current Guidelines from the American College of Rheumatology (ACR), Osteoarthritis Research Society International (OARSI) and the European League against Rheumatism (EULAR) recommend the use of IA corticosteroids for short-term acute pain relief (Hochberg et al, 2012; Jordan et al, 2003; Menge et al, 2014).

The prevalence of hip osteoarthritis is estimated to range from 6.7% to 9.2% among adults ≥45 years of age and increases with age (Lawrence et al, 2008; Murphy et al, 2012). It is recognized that chronic inflammation occurs in all stages of OA (Benito et al, 2005; Sellam and Berenbaum, 2010; Wenham and Conaghan, 2010). As inflammation is correlated with clinical symptoms and joint degeneration, it should be an important target for corticosteroid intervention.

FX006 is an extended-release formulation of triamcinolone acetonide (TA) for IA administration. It is approved in the US under the trade name ZILRETTA® (triamcinolone acetonide extended-release injectable suspension) for the management of pain of osteoarthritis of the knee. FX006 is intended to deliver TA to the synovial and peri-synovial tissues for a period of approximately 3 months (Bodick et al, 2013). FX006 contains TA, United States Pharmacopeia (Ph. Eur/USP), formulated in 75:25 poly (lactic-co-glycolic acid) (PLGA) microspheres with a nominal drug load of 25% (weight by weight [w/w]) and is provided as a sterile white to off-white powder for reconstitution. The drug product is reconstituted with diluent containing an isotonic, sterile aqueous solution of sodium chloride (NaCl; 0.9% w/w), carboxymethylcellulose sodium (CMC; 0.5% w/w) and polysorbate-80 (0.1% w/w) to form a suspension prior to IA injection.

Similar as in knee OA, hip OA patients are confronted with insufficient management of their symptoms (Zhang et al, 2008). Conventional corticosteroids have demonstrated clinical benefits in patients with hip OA (Lambert et al, 2007; Qvistgaard et al, 2006; Atchia et al, 2011), but with short duration of effect (approximately 4-8 weeks) and side effects from burst release of steroids into systemic circulation (Habib et al, 2011). Due to its slow release formulation, FX006 has the potential to offer longer duration of efficacy and minimized systemic exposure, thus, an improved benefit/risk profile for hip OA patients.

Intra-articular administration of FX006, an extended-release microsphere formulation of triamcinolone acetonide, demonstrated safety and efficacy in the relief of pain in patients with pain associated with OA of the knee. Given the insufficient symptomatic management of hip OA patients and similar pathogenesis between knee and hip OA, it is anticipated that FX006 will provide similar benefit to these

Flexion Therapeutics Protocol FX006-2019-017 SAP, Version 1.0 18 December 2019

patients. However, to fully assess the safety, efficacy and determine a benefit/risk profile for administration of FX006 to patients with hip OA, the procedure for IA administration of FX006 into the hip joint needs to be addressed. Thus, the sponsor is proposing a specific study to evaluate the ability of injection procedures to achieve successful IA injection of FX006 into the hip joints of patients with OA of the hip.

### 1.2. Objectives of Statistical Analysis

### Primary:

• To evaluate the ability of injection procedures to achieve successful IA injection of FX006 into the hip joints of patients with OA of the hip.

### Secondary:

• The secondary objective of this study is to assess the safety of FX006 administered by IA injection in patients with hip OA.

This statistical analysis plan (SAP) is designed to outline the methods to be used in the analysis of study data in order to answer the study objective(s). Populations for analysis, data handling rules, statistical methods, and formats for data presentation are provided. The statistical analyses and summary tabulations described in this SAP will provide the basis for the results sections of the clinical study report (CSR) for this trial, as well as be used for regulatory filings and manuscripts and presentations.

This SAP will also outline any differences in the currently planned analytical objectives relative to those planned in the study protocol.

### 2. STUDY DESIGN

### 2.1. Synopsis of Study Design

This is a prospective, multicenter, single-arm, open-label study to evaluate and confirm feasibility of an IA injection procedure of 32 mg FX006 under image guidance in patients with hip OA. The study will be conducted at up to 6 sites with approximately 22 patients. If one (1) unsuccessful IA administration is observed, 7 additional patients may be enrolled. Eligible patients will be administered a single IA injection of FX006 on Day 1 and then followed for safety for 8 weeks.

### 2.2. Study Procedures

Patients participating in this study will complete visit schedules and procedures as detailed in the Schedule of Study Assessments (<u>Table 1</u>).

 Table 1
 Schedule of Study Assessments

| List of Assessments | Screening <sup>1</sup> | Day 1 | Week 1 | Week 4 | Week 8 |
|---|---|---|---|---|---|
| Window | -14 to -1 | _ | ±2 days | ±5 days | ±5 days |
| Informed consent | X | | | | |
| Inclusion/Exclusion Review | X | $X^2$ | | | |
| Medical History/Update | X | $X^2$ | | | |
| Patient Demographics | X | | | | |
| OA Medical History | X | | | | |
| Prior Treatments and<br>Medications | X | $X^2$ | | | |
| Physical examination | X | | | | |
| Vital signs | X | $X^2$ | X | | X |
| Height | X | | | | |
| Weight and BMI | X | | | | |
| Index Hip Assessment | X | $X^2$ | X | | X |
| Index Hip X-ray <sup>3</sup> | X | | | | |
| Hematology, Chemistry <sup>4</sup> | X | | | | |
| HIV, Hep B/C <sup>4</sup> | X | | | | |
| Pregnancy Test <sup>5</sup> | X <sup>5</sup> | $X^{2,5}$ | | | |
| Index Hip Aspiration <sup>6</sup> | | X | | | |
| IP administration <sup>7</sup> | | X | | | |
| AE/SAE & ConMeds <sup>8</sup> | X | X | X | X <sup>9</sup> | X |

<sup>1</sup> Screening period is up to 14 days.

### 2.3. Efficacy Endpoints

### 2.3.1. Primary Efficacy Endpoint

The primary endpoint for this study is successful study drug administration, defined as the Injector reporting the complete administration of study drug.

<sup>2</sup> To be completed on Day 1 prior to injection procedure

<sup>3</sup> A weight-bearing anterior-posterior view for index hip is recommended. Screening X-ray will be read locally for radiologic findings of OA meeting criteria for Kellgren-Lawrence Grade 2-3.

<sup>4</sup> To be performed via local laboratory.

<sup>5</sup> Pregnancy test will be done in women of childbearing potential. Serum Pregnancy Test to be performed at Screening visit by local lab; Urine Pregnancy Test to be performed on Day 1 by study site or local lab with result available prior to injection of study medication.

<sup>6</sup> Aspiration must be attempted prior to IP administration. Synovial fluid volume aspirated will be recorded prior to discard.

<sup>7</sup> To be performed under image guidance in compliance with protocol specified procedure.

<sup>8</sup> AE/SAE's and concomitant medications will be captured from signing of informed consent through EOS visit.

<sup>9</sup> To be conducted via telephone

# 3. PATIENT POPULATIONS

# 3.1. Population Definitions

The following patient populations will be used for presentation and analysis of the data:

• Safety Population: All patients who received an attempted administration of study drug.

### 4. STATISTICAL METHODS

### 4.1. Sample Size Justification

Approximately 22 patients will be treated in this study. If there are no incomplete IA administrations, the study may be considered complete. Observing 0 incomplete injections (0%) in 22 patients gives 90% confidence that the true incomplete IA injection rate is between 0 and 10%. If one (1) unsuccessful IA administration of study drug is observed, 7 additional patients may be enrolled. Observing 1 incomplete IA injection in 29 patients (3%) gives 80% confidence that the true incomplete IA injection rate is between 0 and 10%.

### 4.2. General Statistical Methods and Data Handling

### 4.2.1. General Methods

All outputs will be incorporated into Portable Document Format (PDF) or Word files, sorted and labeled according to the International Conference on Harmonization (ICH) recommendations, and formatted to the appropriate page size(s).

Tables will be presented by a single treatment arm. For categorical variables, summary tabulations of the number and percentage within each category (with a category for missing data) of the parameter will be presented. For continuous variables, the number of non-missing values (n), the mean, median, standard deviation (SD), minimum and maximum values will be presented. 95% confidence intervals (CI) may be provided. Additional statistics may be presented for certain endpoints as described below.

All collected data for enrolled patients will be presented in by-patient listings sorted by patient number. All data listings that contain an evaluation date will contain a relative study day (Rel Day Dose 1). Pretreatment and post-treatment study days are numbered relative to the day of the first dose of study treatment, which is designated as Day 1. The preceding day is Day -1, the day before that is Day -2, etc.

The sections below describe the intended analysis of the endpoints. Additional sensitivity analyses may be employed in the event of any unforeseen data anomalies or data issues not known at the time of writing this analysis plan.

### **4.2.2.** Computing Environment

All descriptive statistical analyses will be performed using SAS® statistical software (Version 9.4 or higher), unless otherwise noted.

Adverse Events (AEs) will be coding using Medical Dictionary for Regulatory Activities (MedDRA) Version 22.0 (or higher).

Concomitant medications will be coded using World Health Organization (WHO) Drug Dictionary (DD) (Version March 1, 2019 or Higher).

### 4.2.3. Methods of Pooling Data

Not applicable to the present study.

### 4.2.4. Adjustments for Covariates

Not applicable to the present study.

### 4.2.5. Multiple Comparisons/Multiplicity

As all analyses are exploratory in nature, there will be no controls for multiplicity.

### 4.2.6. Subpopulations

Analysis of the primary endpoint would be carried out for subgroups defined by aspiration status, KL grade at baseline, and gender.

### 4.2.7. Discontinuations and Loss to Follow-up

Each treated patient from this study receives study medication as a single IA injection. Therefore, discontinuation from treatment is not applicable.

Each patient may only discontinue from the study for further assessments and study visits. Data collected from discontinued patients will be included in the CSR. Patients who discontinue from the study may be replaced at the discretion of the sponsor.

### 4.2.8. Missing, Unused, and Spurious Data

Missing values will not be imputed and data will be analyzed "as observed".

### 4.2.9. Visit Windows

Data collected at unscheduled visits will be mapped to the closest scheduled visit, but only if that data is not already available in that visit. Otherwise data will be summarized and presented according to the nominal visit as recorded on the Electronic Case Report Form (eCRF).

### 4.2.10. Baseline definitions

Baseline is the Baseline/Day 1 assessment prior to administration of the first dose of study treatment. If the Baseline result is missing, the last non-missing result prior to administration of study treatment may be used from the screening period.

### 4.3. Interim Analyses

There will be no interim analyses for this study.

### 4.4. Final Analyses

The analyses of study data will be performed in an unblinded manner when all patients have completed, withdrawn or discontinued from the study. Final analyses specified in the protocol and SAP will be completed and reported in the CSR.

Post-hoc, exploratory analyses, may be completed to further understand and elucidate study results. Any post-hoc, exploratory analyses completed will be clearly identified as such in the final CSR.

### 4.5. Patient Disposition

Patient disposition will be tabulated and include the total number of patients enrolled, treated, completed and early terminated, reason for early termination and the number in each patient population.

The following by-patient data listings will be presented:

- Study completion information including the reason for premature study discontinuation, if applicable.
- Inclusion/exclusion criteria not met.
- Patient inclusion in the Safety Population.

### 4.6. Protocol Deviations

The number and percentage of patients with at least one protocol deviation will be summarized for the Safety Population. Additionally, incidence by type of deviation will be presented in the following categories: inclusion criteria not met, exclusion criteria met, informed consent form (ICF) related, visit out of window, study drug administration, missed visit, missed assessment / procedure, assessment out of window, prohibited medication taken, incorrect assessment sequence / timing, incorrect delegation, documentation issue, and other. In these tabulations, patients could be counted in more than one category if they have a deviation attributed to multiple categories. All protocol deviations will be presented in a data listing.

### 4.7. Demographic and Baseline Characteristics

Demographic and baseline characteristics will be listed by study site and patient and will be summarized. Frequencies and proportions will be presented for the categorical variables and descriptive statistics will be presented for continuous variables.

### 4.7.1. Demographic Characteristics

The following Baseline parameters will be summarized for the Safety Population:

- Age (year) at consent Age will be calculated as the years between date of birth and date of informed consent, and will be rounded down to the nearest year.
- Weight (kilogram (kg));
- Height (centimeter (cm));
- Gender (Male/Female);
- Body mass index (BMI) (kg/meter (m)<sup>2</sup>);
- BMI category:
  - o Underweight: <18.5 kg/m<sup>2</sup>
  - o Normal:  $18.5 \text{ to } < 25.0 \text{ kg/m}^2$
  - $\circ$  Overweight: 25.0 to  $<30.0 \text{ kg/m}^2$
  - Obesity Class I: 30.0 to <35.0 kg/m<sup>2</sup>
  - Obesity Class II: 35.0 to <40.0 kg/m<sup>2</sup>
  - o Obesity Class III: >=40.0 kg/m<sup>2</sup>
- Ethnicity (Hispanic or Latino / Not Hispanic or Latino);
- Race (White / Asian / Black or African American / American Indian or Alaska Native / Native Hawaiian or Other Pacific Islander);
- Age, height, weight, and BMI will be summarized using descriptive statistics (number of patients, mean, SD, median, minimum, and maximum). The number and percentage of patients in each gender, ethnicity, race and BMI category will also be presented.

### **4.7.2. OA Medical History**

OA history and index hip characteristics as collected on the eCRF will be summarized for the SP.

Time from primary diagnosis of OA in the index hip to Day 1 of the study in days (first dose date – date of diagnosis + 1), will be computed and presented descriptively. If only month and year of initial diagnosis is available, day will be imputed as 1 for calculations. If month and day are missing, the time from primary diagnosis will be computed as year of first dose minus year of diagnosis. If year is missing, time from diagnosis will not be computed.

### 4.7.3. Prior medication

All prior medications will be presented in the concomitant medication data listing with a flag identifying which medications are prior medications (refer to Section 4.10.6 for details on defining prior and concomitant medications).

### 4.8. Study Drug Exposure

Details of study drug administration will be summarized for the SP.

Descriptive statistics summarizing the index hip injected, approach for injection, needle size used, numbing agent used, use of fluoroscopy guidance, use of contrast dye or air used to confirm IA placement, total prepared volume, volume injected in the hip joint, air volume injected into hip joint, positioning of patient and index leg/hip, index leg rotation, degrees of rotation, use of connector for FX006 injection, and horizontal positioning of syringe during injection with FX006 will be presented in a summary table.

All study drug exposure data will be presented in a data listing.

### 4.9. Efficacy Evaluation

All efficacy analyses will be conducted using the SP. The rate and 90% CI of successful FX006 administration will calculated using all patients dosed, using methodology for estimation of a binomial proportion. Confidence intervals will be calculated via the score method, including a continuity correction.

Exploratory analyses may be conducted to aid in determination of root causes of unsuccessful injections, should any occur.

In addition to the analyses described above, subgroup analyses will be performed for subgroups defined by aspiration status, KL grade at baseline, and gender.

### 4.10. Safety Analyses

Safety analyses will be conducted using the SP.

### 4.10.1. Adverse Events

AEs will be coded using MedDRA and displayed in tables and listings using System Organ Class (SOC) and Preferred Term (PT).

Analyses of AEs will be performed for those events that are considered treatment emergent, where treatment emergent is defined as any AE with onset after the administration of study treatment, or any event that was present at Baseline but worsened in intensity through the end of the study.

• If the start date/time of an AE is partially or completely missing, the date/time will be compared as far as possible with the date/time of the start of administration of study drug. The AE will be assumed to be treatment emergent if it cannot be definitively shown that the AE did not occur or worsen during the treatment-emergent period (worst case approach). The following general rules will be used:

- If the start time of an AE is missing but the start date is complete, an AE will only be excluded as being treatment emergent if the start date is before the date of study drug administration or if the stop date/time is before study drug administration.
- If the start time and day are missing but the start month and year are complete, an AE will only be excluded as being treatment emergent if the start month/year is before the month/year of study drug administration or if the stop date/time is before study drug administration.
- If the start day and month are missing but the start year is complete, an AE will only be excluded as being treatment emergent if start year is before the year of study drug administration or if the stop date/time is before study drug administration.
- If the start date is completely missing, an AE will be considered treatment-emergent unless the stop date/time is before study drug administration.

AEs will be summarized by patient incidence rates; therefore, in any tabulation, a patient contributes only once to the count for a given SOC or PT.

Summary tables will display the number and percentage of patients who experienced at least one treatment emergent AE (TEAE) in each of the following categories:

- Any TEAE
- Any Serious AE (SAE)
- Any TEAE leading to study discontinuation
- Any TEAE by severity (Mild/Moderate/Severe)
- Any TEAE by relationship
- Any index hip related TEAE
- Any index hip related SAE
- Any index hip related TEAE leading to study discontinuation
- Any index hip related TEAE by severity (Mild/Moderate/Severe)
- Any index hip related TEAE by relationship
- Any TEAE related to injection procedure

Separate tabulations will be produced for each of following categories:

- All TEAEs by SOC and PT
- All TEAEs by PT (decreasing frequency)
- All SAEs by SOC and PT
- All TEAEs related to study drug by SOC and PT
- All TEAEs related to injection procedure by SOC and PT
- All TEAEs by maximum severity by SOC and PT
- All TEAEs leading to study discontinuation by SOC and PT
- All TEAEs leading to death by SOC and PT
- All index hip related TEAEs by SOC and PT
- All index hip related TEAEs related to study drug by SOC and PT
- All index hip related TEAEs by maximum severity by SOC and PT

In the summary table for "Any TEAE by SOC and PT", an additional row with the number of events observed will be presented. A patient will be counted once for the number of patients if they have multiple events. The total number of events will be the absolute number of events observed, and a patient will be counted more than once for the event totals if they have multiple events.

In these tabulations, related is defined as any TEAE deemed related to study drug by the investigator. If relationship is missing, it will be imputed as related.

If an event has a TEAE start date that, after imputation rules are applied, is not complete enough to determine the time period in which the TEAE occurred, that event will not be included in the tabulations by study day.

Formal hypothesis-testing of AE incidence rates will not be performed.

By-patient listings of all AEs occurring on-study will be provided as well as for the following, for all patients: patient deaths, SAEs and AEs leading to discontinuation.

### 4.10.2. Laboratory Data

The Baseline (Screening) values will be summarized for each hematology and clinical chemistry laboratory parameter. All laboratory data, including Common Terminology Criteria for Adverse Events (CTCAE) 4.03 grade, will be provided in data listings. See Section 7.3 for CTCAE grade definitions.

### 4.10.3. Vital Signs and Physical Examinations

The observed value and change from Baseline at Week 1 and Week 8 for vital sign data will be summarized in a summary table. Vital sign measurements include blood pressure, heart rate, oral temperature, and weight, and BMI. Vital sign measurements will be presented for each patient in a data listing.

All physical examination results will be presented in a data listing.

### 4.10.4. Index Hip Assessment and Aspiration

The index hip will be assessed for evidence of inflammation, including tenderness, warmth, redness, swelling, and effusion, limitation on range of motion (directions: flexion, extension, abduction, adduction, internal rotation or external rotation; severity: mild, moderate or severe). Clinically significant findings will be summarized. Index hip assessment data will be presented in a data listing.

Aspiration of the index hip joint must be attempted prior to injection of contrast and study medication at Day 1. The synovial fluid volume, if any, will be measured. Data regarding protocol-required aspiration that is performed at the time of injection in will be included in the summary table and listing for Study Drug Exposure. Additional aspirations, not required per protocol, will be presented in a separate aspiration listing.

### **4.10.5. Index Hip X-Ray**

Index hip X-rays are performed at Screening. The Screening X-ray will be read locally for Kellgren-Lawrence (KL) grading. KL grading at baseline will be summarized, based on the following grades:

- Grade 0: Normal appearance.
- Grade 1: Possible osteophytes, possible Joint Space Narrowing (JSN) medially.
- Grade 2: Definite osteophytes, definite JSN, slight sclerosis.
- Grade 3: Mild osteophytes, marked JSN, moderate sclerosis, cysts and deformity
- Grade 4: Large osteophytes, severe JSN, cysts sclerosis and deformity

A patient listing of index hip X-ray will also be presented.

### 4.10.6. Concomitant Medications

Concomitant medications (CM) will be defined as those medications that were initiated after study drug administration or those that were ongoing at the time of study drug administration. If the start date or stop date of a medication is partially missing, the date will be compared as far as possible with the date of the start of administration of study drug. The medication will be assumed to be prior medication if it cannot be definitively shown that the medication did not start or continue after study drug administration and was not ongoing at the time of study drug administration. The following approach will be taken:

- If the start date of medication is complete and occurs on or after the day of administration of study treatment, the medication will be assumed concomitant. If the start date occurs prior to administration of study treatment but the end date is on or after the administration of study treatment date or the medication is recorded as ongoing, the medication will be considered concomitant.
- If the start day is missing but the start month and year are complete, a medication will only be excluded as being concomitant if the start month/year is before the month/year of study drug administration and if the stop date (either full date, month and year if missing day, or year if missing month and day) is before study drug administration.
- If the start day and month are missing but the start year is complete, a medication will only be excluded as concomitant if the start year is before the year of study drug administration and if the stop date (either full date, month and year if missing day, or year if missing month and day) is before study drug administration.
- If the start date is completely missing and the stop date is prior to administration of study treatment or completely missing, the medication will be assumed to be a prior medication.

All prior and CMs will be presented in a data listing with flags indicating whether each medication was prior and/or concomitant. The listings will include type of medication (general or restrictive) and whether the CM was used for treatment of an AE.

### 4.10.7. Surgical Procedures

Surgical procedures that occurred during the study will be provided in a data listing.

# 5. CHANGES TO PLANNED ANALYSES

| There are no major changes to the planned analyses. |
|-----------------------------------------------------|

### 6. REFERENCES

Atchia I, Kane D, Reed MR, Isaacs JD, Birrell F. Efficacy of a single ultrasound-guided injection for the treatment of hip osteoarthritis. Ann Rheum Dis. 2011 Jan;70(1):110-6.

Benito MJ, Veale DJ, FitzGerald O, van den Berg WB, Bresnihan B. Synovial tissue inflammation in early and late osteoarthritis. Ann Rheum Dis. 2005 Sep;64(9):1263-7.

Bodick N, Lufkin J, Willwerth C, Blanks R, Inderjeeth C, Kumar A, Clayman M. FX006 prolongs the residency of triamcinolone acetonide in the synovial tissues of patients with knee osteoarthritis. Osteoarthritis Cartilage. 2013;21:(Suppl); S144-5.

Cisternas MG, Murphy L, Sacks JJ, Solomon DH, Pasta DJ, Helmick CG. Alternative Methods for Defining Osteoarthritis and the Impact on Estimating Prevalence in a US Population-Based Survey. Arthritis Care Res (Hoboken). 2016;68(5):574–80.

Creamer P, Hochberg MC. Osteoarthritis. Lancet 1997;350(906):503-508.

Goldring SR and Goldring MB. Clinical aspects, pathology and pathophysiology of osteoarthritis. J Musculoskelet Neuronal Interact 2006;6(4):376–378.

Guy W. ECDEU assessment manual for psychopharmacology (DHEW Publication No. ADM 76-338). Washington, DC: US Government Printing Office; 1976.

Habib GS and Miari W. The effect of intra-articular triamcinolone preparations on blood glucose levels in diabetic patients: a controlled study. J Clin Rheumatol 2011;17:302-305.

Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, et al. American College of Rheumatology 2012: Recommendations for the Use of Nonpharmacologic and Pharmacologic Therapies in Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken) 2012; 64(4):465-474.

Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, et al. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis 2003;62(12):1145–1155.

Lambert RG, Hutchings EJ, Grace MG, Jhangri GS, Conner-Spady B, Maksymowych WP. Steroid injection for osteoarthritis of the hip: a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2007 Jul;56(7):2278-87.

Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, et al. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum 2008;58:26-35.

Menge TJ, Boykin RE, Byram IR, Bushnell BD. A Comprehensive Approach to Glenohumeral Arthritis. South Med J. 2014;107(9):567-573.

Flexion Therapeutics Protocol FX006-2019-017 SAP, Version 1.0 18 December 2019

Murphy L, Helmick CG. The impact of osteoarthritis in the United States: a population-health perspective: A population-based review of the fourth most common cause of hospitalization in U.S. adults. Orthop Nurs 2012;31:85-91.

Qvistgaard E, Christensen R, Torp-Pedersen S, Bliddal H. Intra-articular treatment of hip osteoarthritis: a randomized trial of hyaluronic acid, corticosteroid, and isotonic saline. Osteoarthritis Cartilage. 2006 Feb;14(2):163-70.

Sellam J and Berenbaum F. The role of synovitis in pathophysiology and clinical symptoms of osteoarthritis. Nat Rev Rheumatol. 2010 Nov;6(11):625-35.

Wenham CY and Conaghan PG. The role of synovitis in osteoarthritis. Ther Adv Musculoskelet Dis. 2010 Dec;2(6):349-59.

Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, et al. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage 2008;16:137-162.

# 7. CLINICAL STUDY REPORT APPENDICES

# 7.1. Statistical Tables and Figures to be Generated

| Table 14.1.1 | Patient Enrollment and Disposition (All Patients) |
|---|---|
| Table 14.1.2 | Demographic and Baseline Characteristics (Safety Population) |
| Table 14.1.3 | Osteoarthritis History and Index Hip Characteristics (Safety Population) |
| Table 14.1.4 | Summary of Protocol Deviations (Safety Population) |
| Table 14.1.5 | Study Drug Exposure Summary (Safety Population) |
| Table 14.2.1.1 | Summary of Successful FX006 Administration (Safety Population) |
| Table 14.2.1.2 | Summary of Successful FX006 Administration by Aspiration Status (Safety Population) |
| Table 14.2.1.3 | Summary of Successful FX006 Administration by KL Grade at Baseline (Safety Population) |
| Table 14.2.1.4 | Summary of Successful FX006 Administration by Gender (Safety Population) |
| Table 14.3.1.1 | Summary of Treatment-Emergent Adverse Events (Safety Population) |
| Table 14.3.1.2 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.3 | Treatment-Emergent Adverse Events by Preferred Term (Safety Population) |
| Table 14.3.1.4 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Related to Study Drug (Safety Population) |
| Table 14.3.1.5 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Related to Injection Procedure (Safety Population) |
| Table 14.3.1.6 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Maximum Severity (Safety Population) |
| Table 14.3.1.7 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term – Leading to Study Discontinuation (Safety Population) |
| Table 14.3.1.8 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term – Leading to Death (Safety Population) |

| Table 14.3.1.9 | Serious Adverse Events by System Organ Class and Preferred Term (Safety Population) |
|---|---|
| Table 14.3.1.10 | Index Hip-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| Table 14.3.1.11 | Index Hip-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term - Related to Study Drug (Safety Population) |
| Table 14.3.1.12 | Index Hip-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Maximum Severity (Safety Population) |
| Table 14.3.2.1 | Patient Listing of Deaths (All Patients) |
| Table 14.3.2.2 | Patient Listing of Serious Adverse Events (All Patients) |
| Table 14.3.2.3 | Patient Listing of Discontinuations Due to Adverse Events (All Patients) |
| Table 14.4.1.1 | Summary of Hematology Parameters at Baseline (Safety Population) |
| Table 14.4.1.2 | Summary of Chemistry Parameters at Baseline (Safety Population) |
| Table 14.4.1.3 | Summary and Change from Baseline for Vital Signs (Safety Population) |
| Table 14.4.2.1 | Summary of Index Hip Assessments (Safety Population) |
| Table 14.4.2.2 | Summary of Index Hip Aspiration (Safety Population) |

# 7.2. Data Listings to be Generated

| Listing 16.2.1 | Patient Disposition |
|--------------------|-------------------------------------------|
| Listing 16.2.2.1 | Inclusion/Exclusion Criteria Not Met |
| Listing 16.2.2.2 | Protocol Deviations |
| Listing 16.2.3 | Analysis Populations |
| Listing 16.2.4.1.1 | Demographics and Baseline Characteristics |
| Listing 16.2.4.2 | Medical History |
| Listing 16.2.4.3 | Medical History - Hip Osteoarthritis |

| Listing 16.2.4.4 | Medical History - Prior Treatment of Hip Osteoarthritis |
|---|---|
| Listing 16.2.4.5 | Medical History - Other Osteoarthritis |
| Listing 16.2.4.6 | Medical History - Other Osteoarthritis Procedures or Surgeries |
| Listing 16.2.4.7 | Screening Index Hip X-Ray/Kellgren-Lawrence Grade |
| Listing 16.2.5.1 | Study Drug Exposure |
| Listing 16.2.6.1.1 | Efficacy Listing |
| Listing 16.2.7.1 | Adverse Events – Sorted By Patient and Onset Date |
| Listing 16.2.7.2 | Adverse Events – Sorted by System Organ Class, Preferred Term, Treatment, Patient, and Onset Date |
| Listing 16.2.7.3 | Adverse Events – Glossary by MedDRA SOC, Preferred Term and Verbatim |
| Listing 16.2.8.1 | Laboratory Assessment – Hematology |
| Listing 16.2.8.2 | Laboratory Assessment – Chemistry |
| Listing 16.2.8.3 | Screening Laboratory Assessments: HIV, Hep B, Hep C, and Urine/Serum Pregnancy Test Results |
| Listing 16.2.9.1 | Vital Signs |
| Listing 16.2.9.2 | Physical Examination Findings |
| Listing 16.2.9.3 | Index Hip Assessment Results |
| Listing 16.2.9.4 | Index Hip Aspiration Results |
| Listing 16.2.9.5 | Index Hip X-Ray Results |
| Listing 16.2.9.6 | Prior and Concomitant Medications |
| Listing 16.2.9.7 | Surgical Procedures |

# 7.3. Laboratory Unit Conversion Factors

| Laboratory Parameter | Original Unit | Conversion Factor | SI Units |
|---|---|---|---|
| Alanine Aminotransferase | IU/L | x 1 | U/I |
| Albumin | g/dl | x 10 | g/l |
| Albumin | mg/dl | x 1/100 | g/l |
| Albumin | umol/l | x 0.069 | g/l |
| Alkaline Phosphatase | mcKat/l | x 1/0.01667 | U/I |
| Alkaline Phosphatase | umol/l | x 1/0.01668 | U/I |
| Alkaline Phosphatase | mU/ml | x 1 | U/I |
| Alkaline Phosphatase | nKat/l | x 1/16.67 | U/I |
| Alkaline Phosphatase | nmol/dl | x 1/1.667 | U/I |
| Alkaline Phosphatase | IU/I | x 1 | U/I |
| Alkaline Phosphatase | UI/I | x 1 | U/I |
| Alpha-foetoprotein | ng/ml | x 1 | mcg/l |
| Arginine test | mg/dl | x 57.4 | umol/l |
| Aspartate Aminotransferase | IU/L | x 1 | U/I |
| Basophils | /mm^3 | x 1/1000 | 10^9/I |
| Basophils | 10^3/micrl | x 1 | 10^9/l |
| Basophils | 10^3/ml | x 1/1000 | 10^9/l |
| Basophils | 10^3/mmc | x 1 | 10^9/I |
| Basophils | 10°3/mm°3 | x1 | 10^9/I |
| Basophils | 10^6/ml | x 1 | 10^9/I |
| Bicarbonate | mEg/l | x 1 | mmol/l |
| Bilirubin (total) | mg/dl | x 1/0.0584671 | umol/l |
| Bilirubin (total) | mg/l | x 1/0.584671 | umol/l |
| Bilirubin (total) | umol/l | x 1/0.504071 | umol/l |
| BUN | mg/dl | x 0.357 | mmol/l |
| Calcium (II) | | x 0.5 | mmol/l |
| Calcium (II) | meq/l | x 1/4.008 | • |
| | mg/dl | · | mmol/l |
| Calcium (II) | mg/l | x 1/40.08 | mmol/l |
| CEA | ng/ml | x 1 | mcg/l |
| Ceruloplasmin | mg/dl | x 10 | mg/l |
| Chloride | mEq/l | x 1 | mmol/l |
| Cholesterol (total) | mg/dl | x 1/38.67 | mmol/l |
| Chorionic Gonadotrophin | mIU/ml | x 1 | IU/I |
| Copper (serum) | mcg/dl | x 0.1574 | umol/l |
| Creatine kinase | mcKat/l | x 1/0.017 | U/I |
| Creatinine | mg/dl | x 1/0.0113119 | umol/l |
| Creatinine | mg/l | x 1/0.113119 | umol/l |
| Creatinine | micrmol/l | x 1 | umol/l |
| DHEA | mcg/l | x 3.467 | nmol/l |
| DHEA-S | mcg/dl | x 0.027 | umol/l |
| DHEA-S | umol/l | x 1/0.027 | umol/l |
| Eosinophils | /mm^3 | x 1/1000 | 10^9/I |
| Eosinophils | 10^3/micrl | x 1 | 10^9/I |
| Eosinophils | 10^3/ml | x 1/1000 | 10^9/l |
| Eosinophils | 10^3/mmc | x 1 | 10^9/l |
| Eosinophils | 10^3/mm^3 | x 1 | 10^9/l |
| Eosinophils | 10^6/ml | x 1 | 10^9/l |
| Estradiol (female) | pg/ml | x 1/0.2724 | pmol/l |
| Ferritin | ng/ml | x 1 | mcg/l |
| Fibrinogen | g/dl | x 29.41 | umol/l |
| FSH (female) | mIU/mI | x 1 | IU/I |
| GGT | U/I | x 1 | IU/I |
| GGT | UI/I | x 1 | IU/I |
| GGT | mckat/l | x 1/0.017 | IU/I |
| GH | ng/ML | x 1 | mcg/l |
| Glucose | mg/% | x 1/18.0157 | mmol/l |
| Glucose | g/l | x 1/0.180157 | mmol/l |
| Giucose | g/1 | V 1/0.100121 | 1111101/1 |

| Glucose | mg/dl | x 1/18.0157 | mmol/l |
|---|---|---|---|
| HBA1C | % total HB | x 100 | % |
| HBA1C | % | x 1/100 | fract of 1 |
| HDL | mg/dl | x 0.0259 | mmol/l |
| Haematocrit | % | x 0.01 | Vol. Fract. |
| Haemoglobin | g/100 ml | x 10 | g/l |
| Haemoglobin | g/dl | x 10 | g/l |
| Haemoglobin | mmol/l | x 16.1145 | g/l |
| IGF-I | ng/ml | x 1 | mcg/l |
| Insulin | mcg/l | x 1/0.00580765 | pmol/l |
| Insulin | mU/I | x 7.175 | pmol/l |
| Insulin | mcU/ml | x 7.175 | pmol/l |
| Iron (III) | mcg/dl | x 1/5.5847 | umol/l |
| LDH | mckat/l | x 1/0.01666 | IU/I |
| LDH | umol/l*s | x 1/0.01667 | IU/I |
| LDH | mmol/l | x 1/16.67 | IU/I |
| LDH | mmol/l*s | x 1/16.67 | IU/I |
| LDH | mymol/l*s | x 1/0.01667 | IU/I |
| LDH | nkat/l | x 1/16.67 | IU/I |
| LDL | mg/dl | x 0.0259 | mmol/l |
| LH (female) | mIU/mI | x 0.0239 | IU/I |
| Lymphocytes | /mm^3 | x 1/1000 | 10/9/1 |
| Lymphocytes | 10^3/micrl | x 1/1000<br>x 1 | 10^9/I |
| Lymphocytes | 10°3/ml | x 1/1000 | 10^9/I |
| Lymphocytes | 10^3/mmc | x 1/1000<br>x 1 | 10^9/I |
| Lymphocytes | 10^3/mm^3 | x 1<br>x 1 | 10^9/I |
| Lymphocytes | 10^6/ml | x 1 | 10^9/I |
| Magnesium (II) | mEq/l | x 0.5 | mmol/l |
| Magnesium (II) | mg/dl | x 1/2.4305 | mmol/l |
| Mean cell volume | mcm^3 | · · | fL |
| Mean cell volume | | x 1<br>x 1 | fL |
| Mean cell volume | micrmc<br>micrm^3 | x 1<br>x 1 | fL |
| Mean cell volume | 10^-15/l | | fL |
| | | x 1 | |
| Mean cell Hb Mean cell Hb conc. | pg/cell<br>% | x 1<br>x 10 | pg/cell |
| Mean cell Hb conc. | g/100 ml | | g/l |
| Mean cell Hb conc. | | x 10 | g/l |
| | g/dl | x 10<br>x 1/1000 | g/l<br>10^9/l |
| Monocytes | /mm^3 | · | 10^9/I |
| Monocytes Monocytes | 10^3/micrl<br>10^3/ml | x 1<br>x 1/1000 | 10^9/I |
| | 10^3/mmc | · ' | 10^9/I |
| Monocytes | 10^3/mm^3 | x 1<br>x 1 | 10^9/I |
| Monocytes Monocytes | 10^6/ml | | 10^9/I |
| | | x 1 | · . |
| Neutrophils | /mm^3<br>10^3/micrl | x 1/1000 | 10^9/l<br>10^9/l |
| Neutrophils | | x 1 | • |
| Neutrophils Neutrophils | 10^3/ml | x 1/1000 | 10^9/l<br>10^9/l |
| | 10^3/mmc | x 1 | |
| Neutrophils | 10^3/mm^3 | x 1 | 10^9/I |
| Neutrophils | 10^6/ml | x 1 | 10^9/I |
| Packed cell volume | 1/I | x 100 | %<br>mmol/l |
| Phosphate | mg/dl | x 1/3.09737 | mmol/l<br>mmol/l |
| Phosphate | mg/l | x 1/30.9737 | , |
| Phosphate | mEq/dl | x 5 | mmol/l |
| Phosphate | mEq/I | x 0.5 | mmol/l |
| Platelets | /mcl | x 1/1000 | 10^9/ |
| Platelets | /mm^3 | x 1/1000 | 10^9/I |
| Platelets | /nl | x 1 | 10^9/I |
| Platelets | /pl | x 1000 | 10^9/I |
| Platelets | 10^12/ | x 1/1000 | 10^9/I |
| Platelets | 10^3/mcl | x 1 | 10^9/l |

| Districts | 1002/ml | v 1/1000 | 10^9/I |
|---|---|---|---|
| Platelets Platelets | 10^3/ml<br>10^3/mm^3 | x 1/1000<br>x 1 | 10^9/I |
| | 10^3/IIII^3 | <b>+</b> | 10^9/I |
| Platelets Platelets | k/mcl | x 1<br>x 1 | 10^9/I |
| | 10^3/micrl | | 10^9/I |
| Platelets | · | x 1 | • |
| Platelets | 10^3/mmc | x 1 | 10^9/I |
| Platelets | 10^6/ml | x 1 | 10^9/I |
| Potassium ion (K) | mEq/l | x 1 | mmol/l |
| Potassium ion (K) | mg/l | x 1/39.098 | mmol/l |
| Prolactin | ng/ml | x 1 | mcg/l |
| Protein (Total) | g/dl | x 10 | g/l |
| Protein (Total) | mg/dl | x 0.01 | g/l |
| Prothrombin | % | x 1/100 | Fract of 1 |
| PT | seconds | x 1 | seconds |
| PTT | seconds | x 1 | seconds |
| RBC | /mcl | x 1/1000 | 10^12/l |
| RBC | /pl | x 1 | 10^12/l |
| RBC | 10^6/mcl | x 1 | 10^12/l |
| RBC | /nl | x 1000 | 10^12/l |
| RBC | 10^6/mm3 | x 1 | 10^12/l |
| RBC | 10^9/I | x 1000 | 10^12/l |
| RBC | T/L | x 1 | 10^12/l |
| RBC | 10^6/micrl | x 1 | 10^12/I |
| RBC | 10^3/ml | x 1000000 | 10^12/ |
| RBC | 10^6/mmc | x 1 | 10^12/I |
| RBC | 10^6/mm^3 | x 1 | 10^12/ |
| SGOT (AST) | mckat/l | x 1/0.01667 | IU/I |
| SGOT (AST) | umol/I*s | x 1/0.01668 | IU/I |
| SGOT (AST) | mmol/l | x 1/16.67 | IU/I |
| SGOT (AST) | mmol/l*s | x 1/16.67 | IU/I |
| SGOT (AST) | nkat/l | x 1/16.67 | IU/I |
| SGOT (AST) | U/I | · | IU/I |
| SGOT (AST) | UI/I | x 1<br>x 1 | IU/I |
| , , | · | | • |
| SGPT (ALT) | U/I<br>UI/I | x 1 | IU/I<br>IU/I |
| SGPT (ALT) | • | x 1 | |
| Sodium ion (Na) | mEq/I | x 1 | mmol/l |
| Sodium ion (Na) | mg/dl | x 1/2.29898 | mmol/l |
| Sodium ion (Na) | g/l | x 1/0.0229898 | mmol/l |
| TBG | mcg/dl | x 12.87 | nmol/l |
| Thyroxin (T4) | mcg/dl | x 1/0.0776874 | nmol/l |
| Thyroxin (T4) | mcg/l | x 1/0.776874 | nmol/l |
| Thyroxin free (fT4) | ng/dl | x 1/0.0776874 | pmol/l |
| Transferrin | mg/dl | x 1/100 | g/l |
| Triglycerides | mg/dl | x 1/88.5445 | mmol/l |
| Triglycerides | g/l | x 1/0.885445 | mmol/l |
| Triiodothyronine (T3) | ng/dl | x 1/65.0976 | nmol/l |
| Triiodothyronine free (fT3) | pg/dl | 'x 1/65.0976 | pmol/l |
| Triiodothyronine Uptake | % | x 1/100 | fract of 1 |
| TSH (thyrotropin) | mcU/ml | 1 | mU/I |
| TT | seconds | x 1 | seconds |
| Urea | mg/dl | x 1/6.00554 | mmol/l |
| Urea | mg/l | x 1/60.0554 | mmol/l |
| Urea | g/l | x 1/0.0600554 | mmol/l |
| Uric acid | mg/dl | x 59.4800 | umol/l |
| Uric acid | mg/l | x 5.9480 | umol/l |
| Uric acid | umol/l | x 1 | umol/l |
| WBC | 10^3/micrl | x 1/1000 | 10^9/I |
| WBC | /mm^3 | x 1/1000 | 10°9/I |
| WBC | /niii 3 | x 1000 | 10^9/I |
| WBC | 10^3/ml | x 1/1000 | 10^9/I |
| WBC | 10,,2/1111 | x 1/1000 | 10.,9/1 |

| WBC | 10^3/mcl | x 1 | 10^9/I |
|-----|-------------|----------|--------|
| WBC | x 10^3/mm^3 | x 1 | 10^9/I |
| WBC | /mcl | x 1/1000 | 10^9/I |
| WBC | 10^3/mmc | x 1 | 10^9/I |
| WBC | 10^6/ml | x 1 | 10^9/I |

# 7.4. Laboratory Normal Ranges

# Site 033:

| Lab Panel | Analyte | Male - LO | Male - HI | Female - LO | Female - HI | Units |
|---|---|---|---|---|---|---|
| Chemistry | Sodium | 133 | 145 | 133 | 145 | mmol/L |
| Chemistry | Potassium | 3.6 | 5.5 | 3.6 | 5.5 | mmol/L |
| Chemistry | Bicarbonate | 21 | 31 | 21 | 31 | meq/mL |
| Chemistry | Chloride | 96 | 110 | 96 | 110 | mmol/L |
| Chemistry | Calcium | 8.5 | 10.4 | 8.5 | 10.4 | mg/dL |
| Chemistry | Total Bilirubin | 0.1 | 1.5 | 0.1 | 1.5 | mg/dL |
| Chemistry | Alkaline Phosphatase | 39 | 117 | 39 | 117 | U/L |
| Chemistry | Alanine Aminotransferase | 0 | 40 | 0 | 40 | U/L |
| Chemistry | Aspartate Aminotransferase | 0 | 37 | 0 | 37 | U/L |
| Chemistry | Blood Urea Nitrogen | 6 | 19 | 6 | 19 | mg/dL |
| Chemistry | Creatinine | 0.5 | 1.2 | 0.5 | 1.2 | mg/dL |
| Chemistry | Uric Acid | 3.4 | 7 | 3.4 | 7 | mg/dL |
| Chemistry | Glucose | 65 | 99 | 65 | 99 | mg/dL |
| Chemistry | Total Protein | 5.9 | 8.4 | 5.9 | 8.4 | g/dL |
| Chemistry | Albumin | 3.2 | 5.1 | 3.2 | 5.1 | g/dL |
| Hematology | Hemoglobin | 14 | 18 | 12 | 16 | g/dL |
| Hematology | Hematocrit | 42 | 52 | 37 | 47 | % |
| Hematology | Erythrocytes count | 4.7 | 6.1 | 4.2 | 5.4 | x 10 <sup>6</sup> / μl |
| Hematology | Mean Cell Volume | 80 | 94 | 81 | 99 | fL |
| Hematology | Leukocytes | 4.8 | 10.8 | 4.8 | 10.8 | x 10³ / μl |
| Hematology | Neutrophils | 40 | 70 | 40 | 70 | % |
| Hematology | Lymphocytes | 17 | 45 | 17 | 45 | % |
| Hematology | Monocytes | 0 | 12 | 0 | 12 | % |
| Hematology | Eosinophils | 0 | 9 | 0 | 9 | % |
| Hematology | Basophils | 0 | 3 | 0 | 3 | |
| Hematology | Platelets | 150 | 400 | 150 | 400 | x 10 <sup>3</sup> / μl |

# Site 053:

| Lab Panel | Analyte | Male - LO | Male - HI | Female - LO | Female - HI | Units |
|---|---|---|---|---|---|---|
| Chemistry | Sodium | 136 | 145 | 136 | 145 | mmol/L |
| Chemistry | Potassium | 3.5 | 5.2 | 3.5 | 5.2 | mmol/L |
| Chemistry | Bicarbonate | 21 | 32 | 21 | 32 | mmol/L |
| Chemistry | Chloride | 98 | 109 | 98 | 109 | mmol/L |
| Chemistry | Calcium | 8.8 | 10.6 | 8.8 | 10.6 | mg/dL |
| Chemistry | Total Bilirubin | 0.3 | 1 | 0.3 | 1 | mg/dL |
| Chemistry | Alkaline Phosphatase | 33 | 125 | 33 | 125 | U/L |
| Chemistry | Alanine Aminotransferase | 7 | 52 | 7 | 52 | U/L |
| Chemistry | Aspartate Aminotransferase | 13 | 39 | 13 | 39 | U/L |
| Chemistry | Blood Urea Nitrogen | 7 | 25 | 7 | 25 | mg/dL |
| Chemistry | Creatinine | 0.6 | 1.3 | 0.6 | 1.3 | mg/dL |
| Chemistry | Uric Acid | 4.4 | 7.6 | 2.3 | 6.6 | mg/dL |
| Chemistry | Glucose | 65 | 99 | 65 | 99 | mg/dL |
| Chemistry | Total Protein | 6.4 | 8.9 | 6.4 | 8.9 | g/dL |
| Chemistry | Albumin | 3.5 | 5.7 | 3.5 | 5.7 | g/dL |
| Hematology | Hemoglobin | 13.7 | 17.5 | 11.2 | 15.7 | g/dL |
| Hematology | Hematocrit | 40.1 | 51 | 34.1 | 44.9 | % |
| Hematology | Erythrocytes count | 4.63 | 6.08 | 3.93 | 5.22 | x 10 <sup>6</sup> / μl |
| Hematology | Mean Cell Volume | 79 | 92.2 | 79.4 | 94.8 | fL |
| Hematology | Leukocytes | 4.23 | 9.07 | 3.98 | 10.04 | x 10 <sup>3</sup> / μl |
| Hematology | Neutrophils | 1780 | 5380 | 1560 | 6130 | Cell/Cmm |
| Hematology | Lymphocytes | 1.32 | 3.57 | 1.18 | 3.74 | x 10 <sup>3</sup> / μl |
| Hematology | Monocytes | 0.3 | 0.82 | 0.24 | 0.86 | x 10 <sup>3</sup> / μl |
| Hematology | Eosinophils | 0.04 | 0.54 | 0.04 | 0.36 | x 10³ / μl |
| Hematology | Basophils | 0.01 | 0.08 | 0.01 | 0.08 | x 10³ / μl |
| Hematology | Platelets | 163 | 337 | 182 | 369 | x 10³ / μl |

# Site 309:

| Lab Panel | Analyte | Male - LO | Male - HI | Female - LO | Female - HI | Units |
|---|---|---|---|---|---|---|
| Chemistry | Sodium | 136 | 145 | 136 | 145 | mmol/L |
| Chemistry | Potassium | 3.4 | 5 | 3.4 | 5 | mmol/L |
| Chemistry | Bicarbonate | 20 | 31 | 20 | 31 | mmol/L |
| Chemistry | Chloride | 98 | 108 | 98 | 108 | mmol/L |
| Chemistry | Calcium | 8.4 | 10.2 | 8.4 | 10.2 | mg/dL |
| Chemistry | Total Bilirubin | 0 | 1.2 | 0 | 1.2 | mg/dL |
| Chemistry | Alkaline Phosphatase | 35 | 129 | 35 | 129 | U/L |
| Chemistry | Alanine Aminotransferase | 21 | 72 | 9 | 52 | U/L |
| Chemistry | Aspartate Aminotransferase | 0 | 40 | 0 | 34 | U/L |
| Chemistry | Blood Urea Nitrogen (17-60 years) | 5 | 22 | 5 | 22 | mg/dL |
| Chemistry | Blood Urea Nitrogen (>60 years) | 5 | 25 | 5 | 25 | mg/dL |
| Chemistry | Creatinine | 0.5 | 1.3 | 0.5 | 1.3 | mg/dL |
| Chemistry | Uric Acid | 3.4 | 8 | 2.4 | 7 | mg/dL |
| Chemistry | Glucose | 70 | 109 | 70 | 109 | mg/dL |
| Chemistry | Total Protein | 6.6 | 8.7 | 6.6 | 8.7 | g/dL |
| Chemistry | Albumin | 3.5 | 5.7 | 3.5 | 5.7 | g/dL |
| Hematology | Hemoglobin | 14 | 17.5 | 13 | 16 | g/dL |
| Hematology | Hematocrit | 38 | 52 | 35 | 47 | % |
| Hematology | Erythrocytes count | 4.5 | 6 | 4 | 5.2 | x 10 <sup>6</sup> / μl |
| Hematology | Mean Cell Volume | 80 | 100 | 80 | 100 | fL |
| Hematology | Leukocytes | 4.5 | 11 | 4.5 | 11 | x 10³ / μl |
| Hematology | Neutrophils | 44 | 77 | 44 | 77 | % |
| Hematology | Lymphocytes | 16 | 44 | 16 | 44 | % |
| Hematology | Monocytes | 5 | 13 | 5 | 13 | % |
| Hematology | Eosinophils | 0 | 8 | 0 | 8 | % |
| Hematology | Basophils | 0 | 3 | 0 | 3 | % |
| Hematology | Platelets | 140 | 400 | 140 | 400 | x 10 <sup>3</sup> / mcl |

# Site 326:

| Lab Panel | Analyte | Male - LO | Male - HI | Female - LO | Female - HI | Units |
|---|---|---|---|---|---|---|
| Chemistry | Sodium | 135 | 145 | 135 | 145 | mmol/L |
| Chemistry | Potassium | 3.5 | 5.3 | 3.5 | 5.3 | mmol/L |
| Chemistry | Bicarbonate | 22 | 31 | 22 | 31 | mmol/L |
| Chemistry | Chloride | 96 | 108 | 96 | 108 | mmol/L |
| Chemistry | Calcium | 8.5 | 10.5 | 8.5 | 10.5 | mg/dL |
| Chemistry | Total Bilirubin | 0.2 | 1 | 0.2 | 1 | mg/dL |
| Chemistry | Alkaline Phosphatase | 45 | 117 | 45 | 117 | U/L |
| Chemistry | Alanine Aminotransferase | 12 | 42 | 12 | 42 | U/L |
| Chemistry | Aspartate Aminotransferase | 15 | 37 | 15 | 37 | U/L |
| Chemistry | Blood Urea Nitrogen | 7 | 23 | 7 | 23 | mg/dL |
| Chemistry | Creatinine | 0.5 | 1.3 | 0.5 | 1.3 | mg/dL |
| Chemistry | Uric Acid | 3.5 | 7.2 | 2.6 | 6 | mg/dL |
| Chemistry | Glucose | 70 | 99 | 70 | 99 | mg/dL |
| Chemistry | Total Protein | 6.4 | 8.2 | 6.4 | 8.2 | g/dL |
| Chemistry | Albumin | 3.4 | 5 | 3.4 | 5 | g/dL |
| Hematology | Hemoglobin | 13 | 17 | 11.5 | 15.5 | g/dL |
| Hematology | Hematocrit | 39 | 50 | 34.5 | 45 | % |
| Hematology | Erythrocytes count | 4.2 | 5.8 | 3.8 | 5.2 | M/uL |
| Hematology | Mean Cell Volume | 80 | 100 | 80 | 100 | fL |
| Hematology | Leukocytes | 3.8 | 10.5 | 3.8 | 10.5 | K/uL |
| Hematology | Neutrophils | 43 | 77 | 43 | 77 | % |
| Hematology | Lymphocytes | 13 | 44 | 13 | 44 | % |
| Hematology | Monocytes | 2 | 14 | 2 | 14 | % |
| Hematology | Eosinophils | 0 | 6 | 0 | 6 | % |
| Hematology | Basophils | 0 | 2 | 0 | 2 | % |
| Hematology | Platelets | 150 | 400 | 150 | 400 | K/uL |

# Site 330:

| Lab Panel | Analyte | Male - LO | Male - HI | Female - LO | Female - HI | Units |
|---|---|---|---|---|---|---|
| Chemistry | Sodium | 134 | 147 | 134 | 147 | mmol/L |
| Chemistry | Potassium | 3.6 | 5.3 | 3.6 | 5.3 | mmol/L |
| Chemistry | Bicarbonate | 19 | 31 | 19 | 31 | mmol/L |
| Chemistry | Chloride | 95 | 108 | 95 | 108 | mmol/L |
| Chemistry | Calcium | 8.8 | 10.4 | 8.8 | 10.4 | mg/dL |
| Chemistry | Total Bilirubin | 0.2 | 1.3 | 0.2 | 1.3 | mg/dL |
| Chemistry | Alkaline Phosphatase | 40 | 140 | 37 | 127 | U/L |
| Chemistry | Alkaline Phosphatase (>50 years) | 40 | 140 | 42 | 146 | U/L |
| Chemistry | Alanine Aminotransferase | 5 | 46 | 5 | 46 | IU/L |
| Chemistry | Aspartate Aminotransferase | 10 | 50 | 10 | 41 | IU/L |
| Chemistry | Blood Urea Nitrogen | 8 | 25 | 8 | 25 | mg/dL |
| Chemistry | Creatinine | 0.6 | 1.5 | 0.6 | 1.4 | mg/dL |
| Chemistry | Uric Acid (13-60) | 3.5 | 8 | 2.2 | 6.5 | mg/dL |
| Chemistry | Uric Acid (>60 years) | 3.5 | 8 | 2.2 | 7 | mg/dL |
| Chemistry | Glucose | 65 | 99 | 65 | 99 | mg/dL |
| Chemistry | Total Protein | 6 | 8 | 6 | 8 | g/dL |
| Chemistry | Albumin (1-50 years) | 3.6 | 5.1 | 3.6 | 5.1 | g/dL |
| Chemistry | Albumin (>50 years) | 3.4 | 4.9 | 3.4 | 3.9 | g/dL |
| Hematology | Hemoglobin | 13 | 18 | 11.5 | 16 | g/dL |
| Hematology | Hematocrit | 35 | 48 | 35 | 48 | % |
| Hematology | Erythrocytes count | 4.3 | 6 | 3.7 | 5.4 | m/mm3 |
| Hematology | Mean Cell Volume | 78 | 100 | 78 | 100 | fL |
| Hematology | Leukocytes | 4 | 11 | 4 | 11 | k/mm3 |
| Hematology | Neutrophils | 1.6 | 9.3 | 1.6 | 9.3 | k/uL |
| Hematology | Lymphocytes | 0.6 | 5.5 | 0.6 | 5.5 | k/uL |
| Hematology | Monocytes | 0.1 | 1.6 | 0.1 | 1.6 | k/uL |
| Hematology | Eosinophils | 0 | 0.7 | 0 | 0.7 | k/uL |
| Hematology | Basophils | 0 | 0.2 | 0 | 0.2 | k/uL |
| Hematology | Platelets | 130 | 450 | 130 | 450 | k/mm3 |

# 7.5. Laboratory Grade Definitions - CTCAE 4.03

| Lab Parameter | Hypo/Hyper | CTCAE Definition | SI Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|---|---|
| Alanine<br>Aminotransferase | Hyper | Alanine Aminotransferase increased | IU/L | >ULN-3xULN | >3-5xULN | >5-20xULN | >20xULN |
| Albumin | Нуро | Hypoalbuminemia | g/L | <lln-30< td=""><td>&lt;30-20</td><td>&lt;20</td><td>-</td></lln-30<> | <30-20 | <20 | - |
| Alkaline Phosphatase | Hyper | Alkaline Phosphatase increased | IU/L | >ULN-<br>2.5xULN | >2.5-5xULN | >5-20xULN | >20xULN |
| Aspartate<br>Aminotransferase | Hyper | Aspartate Aminotransferase increased | IU/L | >ULN-3xULN | >3-5xULN | >5-20xULN | >20xULN |
| Bilirubin | Hyper | Blood bilirubin increased | umol/L | >ULN-<br>1.5xULN | >1.5-3xULN | >3-10xULN | >10xULN |
| Calcium | Нуро | Hypocalcemia | mmol/L | <lln-2< td=""><td>&lt;2-1.75</td><td>&lt;1.75-1.5</td><td>&lt;1.5</td></lln-2<> | <2-1.75 | <1.75-1.5 | <1.5 |
| Calcium | Hyper | Hypercalcemia | mmol/L | >ULN-2.9 | >2.9-3.1 | >3.1-3.4 | >3.4 |
| Cholesterol | Hyper | Hypercholesterolemia | mmol/L | >ULN-7.75 | >7.75-10.34 | >10.34-12.92 | >12.92 |
| Creatinine | Hyper | Creatinine increased | umol/L | >1-1.5x<br>Baseline; | >1.5-3x<br>Baseline;<br>>1.5-3x ULN | >3x Baseline;<br>>3-6xULN | >6xULN |

| Lab Parameter | Hypo/Hyper | CTCAE Definition | SI Unit | Grade 1<br>>ULN-<br>1.5xULN | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|---|---|
| Glucose Phosphate | Нурег | Hyperglycemia Hypophosphatemia | mmol/L | >ULN-8.9<br><lln-0.8< td=""><td>&gt;8.9-13.9<br/>&lt;0.8-0.6</td><td>&gt;13.9-27.8<br/>&lt;0.6-0.3</td><td>&gt;27.8</td></lln-0.8<> | >8.9-13.9<br><0.8-0.6 | >13.9-27.8<br><0.6-0.3 | >27.8 |
| Potassium | Нуро | Hypokalemia | mmol/L | <lln-3< td=""><td><lln-3< td=""><td>&lt;3-2.5</td><td>&lt;2.5</td></lln-3<></td></lln-3<> | <lln-3< td=""><td>&lt;3-2.5</td><td>&lt;2.5</td></lln-3<> | <3-2.5 | <2.5 |
| Potassium<br>Sodium | Нурег | Hyperkalemia Hyponatremia | mmol/L | >ULN-5.5<br><lln-130< td=""><td>&gt;5.5-6</td><td>&gt;6-7<br/>&lt;130-120</td><td>&gt;7<br/>&lt;120</td></lln-130<> | >5.5-6 | >6-7<br><130-120 | >7<br><120 |
| Sodium<br>Triglycerides | Hyper<br>Hyper | Hypernatremia Hypertriglyceridemia | mmol/L | ULN-150<br>150-300 | >150-155<br>>300-500 | >155-160<br>>500-1000 | >160<br>>1000 |
| Hemoglobin Hemoglobin | Hypo<br>Hyper | Anemia Hemoglobin increased | g/L<br>g/L | <lln-100 in="" increase="">0- 20 above ULN or above Baseline if Baseline is above ULN</lln-100> | <100-80 Increase in >20-40 above ULN or above Baseline if Baseline is above ULN | <80 Increase in >40 above ULN or above Baseline if Baseline is above ULN | - |
| Leukocytes | Нуро | White blood cells decreased | 10^9/L | <lln-3.0< td=""><td>&lt;3.0-2.0</td><td>&lt;2.0-1.0</td><td>&lt;1.0</td></lln-3.0<> | <3.0-2.0 | <2.0-1.0 | <1.0 |

| Lab Parameter | Hypo/Hyper | CTCAE Definition | SI Unit | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|---|---|
| Leukocytes | Hyper | Leukocytosis | 10^9/L | - | - | >100 | - |
| Lymphocytes | Нуро | Lymphocyte count decreased | 10^9/L | <lln-0.8< td=""><td>&lt;0.8-0.5</td><td>&lt;0.5-0.2</td><td>&lt;0.2</td></lln-0.8<> | <0.8-0.5 | <0.5-0.2 | <0.2 |
| Lymphocytes | Hyper | Lymphocyte count increased | 10^9/L | _ | >4-20 | >20 | _ |
| Neutrophils | Нуро | Neutrophils count decreased | 10^9/L | <lln-1.5< td=""><td>&lt;1.5-1</td><td>&lt;1-0.5</td><td>&lt;0.5</td></lln-1.5<> | <1.5-1 | <1-0.5 | <0.5 |
| Platelets | Нуро | Platelet count decreased | 10^9/L | <lln-75< td=""><td>&lt;75-50</td><td>&lt;50-25</td><td>&lt;25</td></lln-75<> | <75-50 | <50-25 | <25 |

The following hematology and chemistry parameters collected in the study are not gradable with CTCAE v4.03:

- Blood Urea Nitrogen
- Bicarbonate (removed from version 4.x; it was available in version 3)
- Chloride
- Erythrocyte Mean Corpuscular Volume
- HDL Cholesterol
- LDL Cholesterol
- Urate
- Basophils
- Eosinophils
- Erythrocytes
- Hematocrit
- Monocytes